CLINICAL TRIAL: NCT02295956
Title: Preoperative Rehabilitation During Neoadjuvant Therapy for Pancreatic Cancer: A Pilot Study
Brief Title: Preoperative Rehabilitation During Neoadjuvant Therapy for Pancreatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0702; NCI-2014-02531 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreatic adenocarcinoma; Preoperative therapy; Questionnaires; Surveys; Exercises; Stretching; Walking; Nutrition counseling; Resistance exercise bands; Phone calls; Booklet; Pamphlet
MeSH Terms: conditions — Pancreatic Neoplasms; Motor Activity | interventions — Surveys and Questionnaires; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Based Exercise and Nutrition Program (Experimental): Series of physical and quality of life assessments administered to participants, taking about 20 minutes to complete. Participants instructed to perform resistance/strengthening exercises for 30 minutes two times each week. Exercise instructional booklet given to all participants describing all exercises. Participants to walk 20-30 minutes at least 3 times a week. Nutrition program discussed with participants. Participants receive phone calls from study staff every 2 weeks for 6 weeks to check for adherence, and if they are having any side effects from the exercise.
  Interventions: Behavioral: Questionnaires; Other: Exercise; Other: Nutrition Counseling; Behavioral: Phone Calls; Other: Booklet

INTERVENTIONS:
Behavioral: Questionnaires — Series of physical and quality of life assessments administered to participants, taking about 20 minutes to complete.
  Other Names: Surveys
Other: Exercise — Participants instructed to perform resistance/strengthening exercises for 30 minutes two times each week. Participants to walk 20-30 minutes at least 3 times a week. Participants issued a set of 3 resistance exercise bands with which the exercises can be performed.
Other: Nutrition Counseling — Within 7 days after being enrolled on study, participant meets with a dietitian to discuss nutrition.
Behavioral: Phone Calls — Participants receive phone calls from study staff every 2 weeks for 6 weeks to check for adherence, and if they are having any side effects from the exercise.
Other: Booklet — Exercise instructional booklet given to all participants describing all exercises.
  Other Names: Pamphlet

SUMMARY:
The goal of this research study is to learn if it is possible to start a home-based exercise and nutrition program for patients with pancreatic cancer or who may have pancreatic cancer before surgery (pre-operative rehabilitation, also known as prehabilitation).

DETAILED DESCRIPTION:
Study Procedures:

If you are found to be eligible to take part in this study, you will be asked to complete additional questionnaires about your physical activity and quality of life. It will take about 20 minutes to complete all of the questionnaires in this study. Your strength and walking speed will also be checked using a hand-held grip test, having you stand from a sitting position five times, and a 6 minute walking test.

The exercise regimen will then be discussed with you. It will include a resistance/ strengthening program and a walking program.

You will receive a booklet and an instructional video describing all of the exercises, a set of resistance tubes and accessories you need to perform all exercises, and a pedometer to count your daily steps. Also, a specialist in rehabilitation along with other study staff will teach you the stretching and strengthening exercises. An MD Anderson rehabilitation doctor will oversee all of this.

Resistance/Strengthening Program:

You will be instructed to perform resistance/strengthening exercises for 30 minutes at least two times each week.

The exercises used in this study are designed to strengthen your muscles. Strengthening certain muscle groups will help with upper body control and balance, which the study staff believes may help with mobility before and after surgery. Also, strengthening the shoulder, back, and leg muscles are important for activities such as getting into and out of bed, which is important after surgeries such as pancreas surgery.

You will be instructed to perform any 8 (out of 19) strengthening exercises for a total of 30 minutes. You will be issued a set of 3 resistance exercise tubes with which the exercises can be performed. The strengthening exercises consist of seated and standing weight-bearing exercises. You will perform 3 sets of 8-12 repetitions each of each exercise. When you are able to perform 3 sets of 12 repetitions of an exercise, you will move up to the next level of resistance (different color tube).

Before the strengthening exercises, you will do a series of 4 standing warm-up exercises that will help with balance.

You will record the date, resistance (color of resistance tube used), number of repetitions and sets, and how hard a session of resistance exercises felt for you. You will also record the total time spent on the strengthening program after each exercise session

You will be encouraged to complete an additional 5 minutes of stretching following the exercises. You will be provided with a handout demonstrating upper body, back, and leg stretches to help prevent soreness.

Walking Program:

The walking program will consist of walking briskly for 20-30 minutes at least 3 times each week. If you are unable to tolerate walking at a brisk speed, you will be instructed to walk at a slower pace. You will be given a pedometer and will be instructed to record the number of steps taken each day in addition to the total time spent during each walking session.

Nutrition:

Within 7 days after being enrolled on this study, you will meet with a dietitian to discuss your nutrition. You will be then be provided with recommendations for calorie, protein, and fluid intake, tools for tracking intake (such as a diet log), as well as goals for weight depending on your treatment/recovery. You will also be instructed to eat a high protein snack/meal/shake within 1 hour after each strengthening session.

Phone Calls:

You will be called every 2 weeks and asked if you are following the exercise and nutrition programs and if you are having any side effects from the exercise (such as pain or difficulty breathing). You will also be asked which resistance band you are using. Each phone call will take about 10-15 minutes.

Length of Study:

You will use the exercise programs during your entire pre-operative period, including during the time you are on other treatments before surgery. In addition, you will continue the exercise program and evaluations for up to 4 months after you have had surgery. If you have a side effect or the disease gets worse, the study staff will decide if continuing the exercise program is in your best interest.

This is an investigational study.

Up to 70 participants will be enrolled on this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pancreatic adenocarcinoma, biopsy-proven or suspected.
2. Scheduled for intended pancreatectomy, > 4 weeks until planned resection.
3. Scheduled for neoadjuvant chemotherapy and/or chemoradiation for pancreatic cancer.
4. Able to understand the description of the study and willing to participate.
5. Able to understand the exercise intervention and able to maintain a daily exercise log.
6. Participant must have telephone access and agree to engage with telephone access with the research personnel.

Exclusion Criteria:

1. Non-English speaking.
2. Unable to complete the baseline assessment questionnaires or functional assessments.
3. Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV).
4. Recent fracture or acute musculoskeletal injury that precludes the ability to weight bear fully on all 4 limbs in order to participate in an exercise intervention.
5. Numeric pain rating scale of >/= 7 out of 10.
6. Myopathic or rheumatologic disease that impacts physical function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Prehabilitation Program Among Pancreatic Patients | 6 weeks
  Feasibility established if > 60% of patients are adherent. Prehabilitation program deemed feasible if 60% or more of participants complete at least 60% of the weekly 150-minute combined walking and strengthening exercises during the 6-week preoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Katz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Houston, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Kurz E, Hirsch CA, Dalton T, Shadaloey SA, Khodadadi-Jamayran A, Miller G, Pareek S, Rajaei H, Mohindroo C, Baydogan S, Ngo-Huang A, Parker N, Katz MHG, Petzel M, Vucic E, McAllister F, Schadler K, Winograd R, Bar-Sagi D. Exercise-induced engagement of the IL-15/IL-15Ralpha axis promotes anti-tumor immunity in pancreatic cancer. Cancer Cell. 2022 Jul 11;40(7):720-737.e5. doi: 10.1016/j.ccell.2022.05.006. Epub 2022 Jun 2. PMID 35660135
- [Derived] Ngo-Huang A, Parker NH, Bruera E, Lee RE, Simpson R, O'Connor DP, Petzel MQB, Fontillas RC, Schadler K, Xiao L, Wang X, Fogelman D, Sahai SK, Lee JE, Basen-Engquist K, Katz MHG. Home-Based Exercise Prehabilitation During Preoperative Treatment for Pancreatic Cancer Is Associated With Improvement in Physical Function and Quality of Life. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419894061. doi: 10.1177/1534735419894061. PMID 31858837
- [Derived] Parker NH, Lee RE, O'Connor DP, Ngo-Huang A, Petzel MQB, Schadler K, Wang X, Xiao L, Fogelman D, Simpson R, Fleming JB, Lee JE, Tzeng CD, Sahai SK, Basen-Engquist K, Katz MHG. Supports and Barriers to Home-Based Physical Activity During Preoperative Treatment of Pancreatic Cancer: A Mixed-Methods Study. J Phys Act Health. 2019 Dec 1;16(12):1113-1122. doi: 10.1123/jpah.2019-0027. Epub 2019 Oct 7. PMID 31592772
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org